CLINICAL TRIAL: NCT00416767
Title: Study of First-Line Therapy Comprising Leucovorin Calcium, Fluorouracil, and Irinotecan (FOLFIRI) in Patients With Progressive Locally Advanced or Metastatic Duodenal-Pancreatic Endocrine Tumors
Brief Title: Combination Chemotherapy as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Neuroendocrine Tumors of the Duodenum or Pancreas That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453858; FFCD-0302; EU-20544; PFIZER-FFCD-0302
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Neoplastic Syndrome
Keywords: metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; recurrent islet cell carcinoma
MeSH Terms: conditions — Adenoma, Islet Cell; Neoplasms; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma; Carcinoma, Islet Cell | interventions — Fluorouracil; Irinotecan; Leucovorin

ARMS (1):
- FOLFIRI (Experimental)
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works as first-line therapy in treating patients with locally advanced or metastatic neuroendocrine tumors of the duodenum or pancreas that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month progression-free survival rate in patients with unresectable locally advanced or metastatic neuroendocrine tumors of the duodenum/pancreas treated with fluorouracil, leucovorin calcium, and irinotecan hydrochloride as first-line chemotherapy.

Secondary

* Determine tumor and biologic response at 6, 12, 18, and 24 months in patients treated with this regimen.
* Determine the duration of response of the primary tumor in patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroendocrine tumor of the duodenum/pancreas by histology or bone scan
* Functional or nonfunctional tumor

  * Tumor meets ≥ 1 of the following criteria:

    * Hepatic or extrahepatic metastases
    * Progressive locally advanced tumor (primary or adenopathies)
* Unresectable disease
* Tumor differentiated and meets the following criteria:

  * Ki 67 ≤ 15%
  * Less than 10 mitoses per 10 large fields
* Measurable or evaluable disease

  * Target lesions must meet 1 of the following criteria within the past 6 months:

    * Increase of 20% in the longest diameter
    * New metastases detected
  * Minimum size of lesions must be 1 of the following:

    * More than 15 mm for metastases
    * More than 50 mm for primary tumor or local lymph nodes

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Creatinine ≤ 1.5 mg/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.8 mg/dL
* No coronary insufficiency or symptomatic cardiac disease
* No intestinal obstruction, enteropathy, or uncontrolled chronic diarrhea
* No Gilbert's disease
* No psychological, social, familial, or geographic condition that would preclude study treatment
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* No other condition that would preclude study therapy

PRIOR CONCURRENT THERAPY:

* No prior adjuvant radiotherapy
* At least 3 months since prior interferon
* Prior somatostatin analogs or antisecretories allowed
* No other prior treatment for this cancer
* No concurrent radiotherapy to the target lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Cadiot, Study Chair — CHU - Robert Debre

REFERENCES:
- [Result] Cadiot G, Bonnetain F, Landi B, et al.: Simplified LV5FU2-irinotecan (FOLFIRI) in the first-line therapy of well-differentiated endocrine carcinomas of the duodeno- pancreatic area: preliminary results of the FFCD 0302 phase II trial with GTE participation. [Abstract] J Clin Oncol 25 (Suppl 18): A-4620, 2007.
- [Result] Brixi-Benmansour H, Jouve JL, Mitry E, Bonnetain F, Landi B, Hentic O, Bedenne L, Cadiot G. Phase II study of first-line FOLFIRI for progressive metastatic well-differentiated pancreatic endocrine carcinoma. Dig Liver Dis. 2011 Nov;43(11):912-6. doi: 10.1016/j.dld.2011.07.001. Epub 2011 Aug 9. PMID 21831734